CLINICAL TRIAL: NCT01375933
Title: A Phase 3, Multicenter, Double-Blinded, Randomized, Study to Assess Comparability of a Single Phase 3 Lot and a Single Commercial Lot of 3'-Aminomethylnicotine-P. Aeruginosa r-Exoprotein A Conjugate Vaccine (NicVAX) in Healthy Adult Smokers
Brief Title: A Comparability Study of the Phase 3 Lot and a Single Commercial Lot of NicVAX in Healthy Adult Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabi-4516
Record Dates: First submitted 2011-06-15; First posted 2011-06-20 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Smoking
Keywords: Smoking; NicVAX; Smoking vaccine
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NicVAX - Phase 3 Lot (Active Comparator): NicVAX - Phase 3 Lot
  Interventions: Biological: NicVAX Vaccine
- NicVAX - Commercial Lot (Active Comparator): NicVAX - Commercial Lot
  Interventions: Biological: NicVAX Vaccine

INTERVENTIONS:
Biological: NicVAX Vaccine — NicVAX Vaccine given 6 times over 6 months

SUMMARY:
The purpose of this study is to assess the comparability of the phase 3 lot and a single commercial lot of NicVAX in healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female smokers, age 18-55, who are currently smoking at least 10 cigarettes per day.

Exclusion Criteria:

* Prior exposure to NicVAX or any other nicotine vaccine.
* History of clinically significant allergic reactions.
* Use of systemic steroids.
* Cancer or cancer treatment within 5 years.
* HIV infection.
* History of drug or alcohol abuse or dependence.
* Required treatment for depression within the past 12 months.
* Body mass index ≥ 30 [calculated as weight (kg)/height2 (m)].
* Significant cardiovascular, hepatic, renal, psychiatric and/or respiratory disease.
* Inability to fulfill all visits for approximately 30 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | At Week 14
  To compare imunogenicity of two lots by serum antibody concentration

SECONDARY OUTCOMES:
Safety | Through Week 16
  Assess safety by adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Nabi Biopharmaceuticals
Locations (6):
- United States (6):
  - NicVAX Investigator, Huntsville, Alabama
  - NicVAX Investigator, San Diego, California
  - NicVAX Investigator, Melbourne, Florida
  - NicVAX Investigator, Peoria, Illinois
  - NicVAX Investigator, South Bend, Indiana
  - NicVAX Investigator, Rockville, Maryland